CLINICAL TRIAL: NCT02008357
Title: Anti-Amyloid Treatment in Asymptomatic Alzheimer's Disease (A4 Study)
Brief Title: Clinical Trial of Solanezumab for Older Individuals Who May be at Risk for Memory Loss
Acronym: A4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15275; H8A-MC-LZAZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Cognition Disorders
Keywords: Cognition; Prevention
MeSH Terms: conditions — Cognition Disorders | interventions — solanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solanezumab/Solanezumab (Experimental): Participants received 400 milligram (mg) solanezumab followed by 800 mg solanezumab and then 1600 milligram solanezumab administered intravenously (IV) every 4 weeks (Q4W) for approximately 240 weeks in double-blind placebo-controlled period.
  Participants begin open label extension and received 1600 mg solanezumab Q4W for 204 weeks (from week 240 to week 444).
  Interventions: Drug: Solanezumab
- Placebo/Solanezumab (Placebo Comparator): Participants received placebo administered IV Q4W for approximately 240 weeks in double-blind period.
  Participants begin open label extension period and received 1600 mg solanezumab Q4W for 204 weeks (from week 240 to week 444).
  Interventions: Drug: Placebo; Drug: Solanezumab

INTERVENTIONS:
Drug: Placebo — Administered IV
  Arms: Placebo/Solanezumab
Drug: Solanezumab — Administered IV
  Other Names: LY2062430

SUMMARY:
The purpose of this study is to test whether an investigational drug called solanezumab can slow the progression of memory problems associated with brain amyloid (protein that forms plaques in the brains of people with Alzheimer Disease [AD]).

DETAILED DESCRIPTION:
The A4 study is a clinical trial for older individuals who have evidence of amyloid plaque build-up in their brains who may be at risk for memory loss and cognitive decline due to Alzheimer's disease. The A4 study will test an anti-amyloid investigational drug in older individuals who do not yet show symptoms of Alzheimer's disease cognitive impairment or dementia with the aim of slowing memory and cognitive decline. The A4 study will also test whether anti-amyloid treatment can delay the progression of AD related brain injury on imaging and other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Has a Mini-Mental State Examination (MMSE) score at screening of 25 to 30
* Has a global Clinical Dementia Rating (CDR) scale score at screening of 0
* Has a Logical Memory II score at screening of 6 to 18
* Has a florbetapir positron emission tomography (PET) scan that shows evidence of brain amyloid pathology at screening
* Has a study partner that is willing to participate as a source of information and has at least weekly contact with the participant (contact can be in-person, via telephone or electronic communication)

Exclusion Criteria:

* Is receiving a prescription acetylcholinesterase inhibitor (AChEI) and/or memantine at screening or baseline
* Lacks good venous access, such that intravenous drug delivery or multiple blood draws would be precluded
* Has current serious or unstable illness including cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic, psychiatric, immunologic, or hematologic disease or other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study
* Has had a history within the last 5 years of a serious infectious disease affecting the brain (including neurosyphilis, meningitis, or encephalitis) or head trauma resulting in protracted loss of consciousness
* Has had a history within the last 5 years of a primary or recurrent malignant disease with the exception of any in situ cancer that was appropriately treated and is being appropriately monitored, such as resected cutaneous squamous cell carcinoma in situ or in situ prostate cancer with normal prostate-specific antigen post-treatment
* Has a known history of human immunodeficiency virus (HIV), clinically significant multiple or severe drug allergies, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, or exfoliative dermatitis)
* Is clinically judged by the investigator to be at serious risk for suicide
* Has a history within the past 2 years of major depression or bipolar disorder as defined by the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM)
* Has a history within the past 5 years of chronic alcohol or drug abuse/dependence as defined by the most current version of the DSM

Open-Label Inclusion Criteria:

* All participants who complete the placebo-controlled period will be allowed to continue into the open-label period

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1169 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (68):
- United States (62):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Health Research Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Institute for Memory Impairment & Neurological Disorders, Irvine, California
  - University of California - San Diego, La Jolla, California
  - University of Southern California School of Medicine, Los Angeles, California
  - University of California - Los Angeles, Los Angeles, California
  - Univ of California Irvine College of Medicine, Orange, California
  - Veterans Affairs Medical Center Palo Alto, Palo Alto, California
  - Sutter Medical Group, Sacramento, California
  - Univ of California San Francisco, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - University of California, Davis - Health Systems, Walnut Creek, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Wien Center for Clinical Research, Miami Beach, Florida
  - Compass Research - Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Compass Research -The Villages, The Villages, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush Alzheimer's Disease Center, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Hospital, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Univ of Nebraska Med Center, Omaha, Nebraska
  - Cleveland Clinic of Las Vegas, Las Vegas, Nevada
  - Dent Neurological Institute, Amherst, New York
  - New York University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Case Western Reserve University, Beachwood, Ohio
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Drexel University College of Medicine at EPPI, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Butler Hospital, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington
  - University of Wisconsin-Madison Hospital and Health Clinic, Madison, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parkville, Victoria, Australia
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
  - Sunnybrook Health Sciences Centre, Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City, Japan

REFERENCES:
- [Derived] Hibar DP, Bauer A, Rabe C, Borlinghaus N, Jethwa A, Kollmorgen G, Di Domenico A, Zetterberg H, Blennow K, Masters CL, Sperling RA, Bittner T. Elecsys pTau217 plasma immunoassay detection of amyloid pathology in clinical cohorts. Alzheimers Dement. 2026 Jan;22(1):e71009. doi: 10.1002/alz.71009. PMID 41537338
- [Derived] Shirzadi Z, Schultz AP, Loghmani N, Yang HS, Ford J, Yaari R, Properzi M, Yau WW, Liu L, Rafii MS, Donohue MC, Brickman AM, Jack CR Jr, Greenberg SM, Aisen P, Sperling RA, Chhatwal JP; A4 Study Team. Independent effects of white matter lesion volume and APOE varepsilon4 on ARIA-H in A4 Study. Alzheimers Dement. 2025 Oct;21(10):e70751. doi: 10.1002/alz.70751. PMID 41085172
- [Derived] Digma LA, Young CB, Winer JR, Cody KA, Younes K, Sheng J, Insel PS, Rissman RA, Sperling R, Mormino EC. Continuum of Core 1 Biomarkers in Preclinical Alzheimer's Disease. medRxiv [Preprint]. 2025 Sep 19:2025.09.17.25336007. doi: 10.1101/2025.09.17.25336007. PMID 41001450
- [Derived] Farina FR, Bennett M, Grill JD, Sperling R, Lawlor B, Griffith JW. Association of Alzheimer's disease concerns with amyloid burden and lifestyle behaviors in cognitively unimpaired older adults. Alzheimers Dement. 2025 Jun;21(6):e70225. doi: 10.1002/alz.70225. PMID 40476544
- [Derived] Dubbelman MA, Liu A, Donohue MC, Langford O, Raman R, Rentz DM, Amariglio R, Sperling RA, Aisen PS, Marshall GA; as the A4 Study team. Changes in Daily Functioning in Association With Tau and Amyloid Among Unimpaired Older Adults With and Without Elevated Amyloid. Neurology. 2025 Jun 24;104(12):e213775. doi: 10.1212/WNL.0000000000213775. Epub 2025 May 29. PMID 40440591
- [Derived] Sperling RA, Donohue MC, Raman R, Rafii MS, Johnson K, Masters CL, van Dyck CH, Iwatsubo T, Marshall GA, Yaari R, Mancini M, Holdridge KC, Case M, Sims JR, Aisen PS; A4 Study Team. Trial of Solanezumab in Preclinical Alzheimer's Disease. N Engl J Med. 2023 Sep 21;389(12):1096-1107. doi: 10.1056/NEJMoa2305032. Epub 2023 Jul 17. PMID 37458272
- [Derived] Lewis CK, Bernstein OM, Grill JD, Gillen DL, Sultzer DL. Anxiety and Depressive Symptoms and Cortical Amyloid-beta Burden in Cognitively Unimpaired Older Adults. J Prev Alzheimers Dis. 2022;9(2):286-296. doi: 10.14283/jpad.2022.13. PMID 35543002
- [Derived] Grober E, Lipton RB, Sperling RA, Papp KV, Johnson KA, Rentz DM, Veroff AE, Aisen PS, Ezzati A. Associations of Stages of Objective Memory Impairment With Amyloid PET and Structural MRI: The A4 Study. Neurology. 2022 Mar 29;98(13):e1327-e1336. doi: 10.1212/WNL.0000000000200046. Epub 2022 Feb 23. PMID 35197359
- See also: A Study of Solanezumab in Older Participants Who May be at Risk for Memory Loss (A4) — https://trials.lillytrialguide.com/en-US/trial/4qngyPbBRKqiYWCI0ouGIQ

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol and statistical analysis plan (SAP), delayed-start analyses were not conducted because no treatment difference was observed at the end of the double-blind (placebo-controlled) period. Hence, data were not evaluated for outcome measure analyses (week 336), but safety data were analyzed for open-label extension period.
Groups:
- Solanezumab/Solanezumab: Participants received 400 milligram (mg) solanezumab followed by 800 mg solanezumab and then 1600 milligram solanezumab administered intravenously (IV) every 4 weeks (Q4W) for approximately 240 weeks in double-blind (placebo-controlled) period.
  Participants begin open label extension period and received 1600 mg solanezumab Q4W for 204 weeks (from week 240 to week 444).
- Placebo/Solanezumab: Participants received placebo administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
  Participants begin open label extension period and received 1600 mg solanezumab Q4W for 204 weeks (from week 240 to week 444).
Period: Double-blind (Placebo Controlled) Period
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Started | 578 | 591
Completed | 406 | 424
Not Completed | 172 | 167
Not completed — Adverse Event | 29 | 35
Not completed — Withdrawal by Subject | 101 | 88
Not completed — Death | 6 | 5
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 3 | 6
Not completed — Coordinating Center Request | 1 | 0
Not completed — Covid-19 Pandemic Disruption | 6 | 3
Not completed — Investigator Recommendation | 2 | 2
Not completed — Non-Compliance | 1 | 1
Not completed — Non-Site Clinician Recommendation | 2 | 0
Not completed — Safety Risk | 2 | 6
Not completed — Started Prohibited Medication | 0 | 1
Not completed — Starting A New Treatment For Alzheimer's Disease | 1 | 1
Not completed — Starting New Trial | 2 | 0
Not completed — Study Partner Unwilling Or Unable To Participate | 3 | 1
Not completed — Family Issues | 1 | 1
Not completed — Subject Relocated to Another Place | 4 | 2
Not completed — Subject's Expectation From Study Were not Aligned | 0 | 3
Not completed — Personal Reason | 0 | 1
Not completed — Discontinued Study due to Health Issues | 3 | 0
Not completed — Site Closure | 0 | 1
Not completed — Medical Health of Study Partner | 0 | 1
Not completed — No Longer Wishes to Participate | 1 | 2
Not completed — Subject Concurrently Enrolled in Another Clinical Drug Trial | 0 | 1
Not completed — Starting Another Treatment for the Disease | 0 | 1
Not completed — Decision was Taken by Subject's Personal Doctor | 1 | 0
Not completed — Inability to have MRI due to Stimulator Implant | 0 | 1
Period: Open-label Extension Period
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Started | 383 (Not all Participants who completed the Double-blind (Placebo Controlled) Period entered into Open-label Extension Period.) | 401 (Not all Participants who completed the Double-blind (Placebo Controlled) Period entered into Open-label Extension Period.)
Completed | 1 | 1
Not Completed | 382 | 400
Not completed — Adverse Event | 8 | 7
Not completed — Death | 7 | 4
Not completed — Lack of Efficacy | 9 | 5
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 27 | 32
Not completed — Study Terminated By Sponsor | 300 | 313
Not completed — Safety Risk | 2 | 1
Not completed — Non-Compliance | 0 | 1
Not completed — Investigator Recommendation | 0 | 1
Not completed — Covid-19 Pandemic Disruption | 0 | 1
Not completed — Coordinating Center Request | 2 | 4
Not completed — No Longer Wishes to Participate | 1 | 1
Not completed — Study Ended | 20 | 25
Not completed — Personal Reasons | 0 | 1
Not completed — Discontinued Study Due to Health Issues | 0 | 2
Not completed — Travel Issues/Limitations | 2 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Solanezumab/Solanezumab: Participants received 400 mg solanezumab followed by 800 mg solanezumab and then 1600 milligram solanezumab administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
  Participants begin open label extension and received 1600 mg solanezumab Q4W for 204 weeks (from week 240 to week 444).
- Total: Total of all reporting groups
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab | Total
Number analyzed (Participants) | 578 | 591 | 1169
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (4.6) | 71.9 (5.0) | 71.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 337 | 357 | 694
  Male | 241 | 234 | 475
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 18 | 34
  Not Hispanic or Latino | 556 | 568 | 1124
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 11 | 13 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 16 | 28
  White | 545 | 555 | 1100
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26 | 22 | 48
  United States | 497 | 513 | 1010
  Japan | 9 | 8 | 17
  Australia | 46 | 48 | 94
Preclinical Alzheimer Cognitive Composite (PACC) Total Score [Mean (Standard Deviation); unit: score on a scale] — PACC has 4 components: Free and Cued Selective Reminding Test (0 (worst)-48 (best recall); Delayed Paragraph Recall test (Range 0 (worst)-25 (best recall); Wechsler Adult Intelligence scale: (ranges 0 [none]-135 [best performance]) and Mini Mental State Examination (Range 0 [worst] - 30 [best performance]). Component scores are transformed using an established normalization method into z-scores. Each of 4 component change scores is divided by baseline sample standard deviation (SD) of that component. Population: PACC z scores are summed to form the composite score. Thus, a change of 1 baseline standard deviation on each component would correspond to a 4-point change on the composite. A z-score of 0 is equal to the mean and implies how many SD higher or lower score as compared with baseline score, with increase signifying improvement. Analysis population description included all randomized participants who had baseline PACC total score data.
  score on a scale
    number analyzed (Participants) | 572 | 591 | 1163
    (all) | 0.01 (2.76) | 0.01 (2.60) | 0.01 (2.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Preclinical Alzheimer Cognitive Composite (PACC) Score
Description: PACC has 4 components: Free and Cued Selective Reminding Test (0 (worst)-96 (best recall); Delayed Paragraph Recall test (Range 0 (worst)-25 (best recall); Wechsler Adult Intelligence scale: Digit Symbol Substitution Test (DSST): (ranges 0 [none]-91 [best performance]) and Mini Mental State Examination (Range 0 [worst] - 30 [best performance]). Component scores are transformed using an established normalization method into z-scores. Each of 4 component change scores is divided by baseline sample standard deviation (SD) of that component. These z scores are summed to form the composite score. Thus, a change of 1 baseline standard deviation on each component would correspond to a 4-point change on the composite. A z-score of 0 is equal to the mean and implies how many SD higher or lower score as compared with baseline score, with increase signifying improvement.
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment. Least square mean (LS) mean was derived using natural cubic spline models with factors for treatment, time, and covariates = age, baseline florbetapir cortical standardized uptake value ratio (SUVr) score, years of education, APOE4 carrier status (n),pacc components version type.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Solanezumab: Participants received 400 mg solanezumab followed by 800 mg solanezumab and then 1600 milligram solanezumab administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
- Placebo: Participants received placebo administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 403 | 426
score on a scale | -1.43 (0.21) | -1.13 (0.16)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Test type: Superiority; p = 0.260, Natural Cubic Spline (NCS) method; LS Mean difference (Final Values) = -0.30, 95% CI 2-sided [-0.816 to 0.220], Standard Error of Mean 0.26

2. Primary Outcome: Change From Baseline of the Preclinical Alzheimer Cognitive Composite (PACC) Score
Description: as for outcome 1
Time Frame: Baseline, Week 336
Population: Zero participants analyzed. Delayed-start analyses were not conducted because no treatment difference was observed at the end of the placebo-controlled period. Hence, data were not evaluated for outcome measure analyses (week 336) in open-label extension period.
Groups:
- Solanezumab/Solanezumab; Placebo/Solanezumab: Participants received 1600 mg solanezumab administered IV Q4W for 204 weeks (from week 240 to week 444) in open-label extension period.
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in Cognitive Function Index (CFI)
Description: The CFI is a modified version of the Mail-in Cognitive Function Screening Instrument, a participant- and study partner/informant-reported outcome measure developed by the Alzheimer's Disease Cooperative Study (ADCS). This assessment includes 15 questions (14 of which contribute to the total score, and 1 additional unscored item) that assess the participant's perceived ability to perform high-level functional tasks in daily-life and sense of overall cognitive functional ability. Study participants and their informants independently rate the participant's abilities. A total score is calculated by combining participant-reported and an informant-reported scores, and ranges from 0 to 14 (yes=1; no=0; maybe=0.5 for each question) with higher scores indicating greater impairment. LS mean was derived using natural cubic spline models with factors for treatment, time, and covariates = age, baseline florbetapir cortical SUVr score, years of education, APOE4 carrier status (n).
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 408 | 422
score on a scale | 1.94 (0.20) | 1.47 (0.20)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Test type: Superiority; p = 0.100, Natural Cubic Spline (NCS) method; LS Mean difference (Final Values) = 0.47, 95% CI 2-sided [-0.089 to 1.020], Standard Error of Mean 0.28

4. Secondary Outcome: Change From Baseline in Cognitive Function Index (CFI)
Description: The CFI is a modified version of the Mail-in Cognitive Function Screening Instrument, a participant- and study partner/informant-reported outcome measure developed by the ADCS. This assessment includes 15 questions (14 of which contribute to the total score, and 1 additional unscored item) that assess the participant's perceived ability to perform high-level functional tasks in daily-life and sense of overall cognitive functional ability. Study participants and their informants independently rate the participant's abilities. A total score is calculated by combining participant-reported and an informant-reported scores, and ranges from 0 to 14 (yes=1; no=0; maybe=0.5 for each question) with higher scores indicating greater impairment.
Time Frame: Baseline, Week 336
Population: as for outcome 2
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities Daily Living-Prevention Questionnaire (ADCS-ADL-Prevention Questionnaire) Score
Description: The ADCS-ADL-prevention questionnaire is a functional measure composed of 18 items that includes 15 activities of daily living rated on a 4-point scale and 3 high level function items. Study participants and their informants independently rate the participant's level of ability (with no difficulty = 3, with some difficulty = 2, with a lot of difficulty = 1, did not do/don't know = 0). Informants are additionally asked to evaluate whether activities were completed less often, required more time to complete, and if any errors were made performing the task. High-level function items are rated as "yes" or "no". The total score is the sum of the scores of the 15 activities of daily living questions (range: 0-45) with higher scores indicating less impairment.
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment. LS mean was derived using natural cubic spline models with factors for treatment, time, and covariates = age, baseline florbetapir cortical SUVr score, years of education, APOE4 carrier status (n).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 408 | 423
score on a scale | -2.29 (0.24) | -1.70 (0.24)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Test type: Superiority; p = 0.082, Natural Cubic Spline (NCS) method; LS Mean difference (Final Values) = -0.59, 95% CI 2-sided [-1.265 to 0.076], Standard Error of Mean 0.34

6. Secondary Outcome: Change From Baseline in Alzheimer's Disease Cooperative Study-Activities Daily Living-Prevention Questionnaire (ADCS-ADL-Prevention Questionnaire) Score
Description: The ADCS-ADL-prevention questionnaire is a functional measure composed of 18 items that includes 15 activities of daily living rated on a 4-point scale and 3 high level function items. Study participants and their informants independently rate the participant's level of ability (with no difficulty = 3, with some difficulty = 2, with a lot of difficulty = 1, did not do/don't know = 0). Informants are additionally asked to evaluate whether activities were completed less often, required more time to complete, and if any errors were made performing the task. High-level function items are rated as "yes" or "no". The scores range from 0 to 45 with higher scores indicating less impairment. The total score is the sum of the scores of the 15 activities of daily living questions (range: 0-45) with higher scores indicating less impairment.
Time Frame: Baseline, Week 336
Population: as for outcome 2
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Mean Composite Standardized Uptake Value Ratio (SUVr)
Description: Deposition of abnormal tau protein in the brain associated with AD was assessed by quantitative positron emission tomography (PET) scan using flortaucipir F-18. Flortaucipir is an F-18-labeled small molecule that binds with high affinity and selectivity to aggregated tau, and provides a measure of aggregated tau deposition in the brain, expressed as flortaucipir SUVr. LS Mean was calculated using an analysis of covariance (ANCOVA) model with fixed effects of baseline florbetapir result, treatment, APOE4 Carrier Status (yes/no), and age at baseline
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: standardized uptake value ratio (SUVr)
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 462 | 477
standardized uptake value ratio (SUVr) | 0.066 (0.0052) | 0.108 (0.0051)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -0.042, 95% CI 2-sided [-0.057 to -0.028], Standard Error of Mean 0.0073

8. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Tau Biomarkers
Description: CSF concentrations of total tau and tau phosphorylated protein concentrations were analyzed using validated Immunoassay method. LS mean was derived using an analysis of covariance (ANCOVA) model with fixed effects of baseline CSF, treatment, APOE4 Carrier Status (yes/no) and age at baseline.
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: nanograms per liter (ng/L)
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 48 | 52
nanograms per liter (ng/L)
  CSF Tau Protein | -17.201 (23.5807) | -20.440 (22.6457)
  CSF Phosphorylated Tau Protein: number analyzed (Participants) | 44 | 46
  CSF Phosphorylated Tau Protein | 10.266 (1.8792) | 11.231 (1.8371)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Cerebrospinal fluid Tau Protein Immunoassay; Test type: Superiority; p = 0.922, ANCOVA; LS Mean difference (Final Values) = 3.239, 95% CI 2-sided [-62.020 to 68.498], Standard Error of Mean 32.8719
Statistical Analysis 2: Comparison: Solanezumab vs Placebo; Cerebrospinal Fluid Phosphorylated Tau Protein Immunoassay; Test type: Superiority; p = 0.717, ANCOVA; LS Mean difference (Final Values) = -0.965, 95% CI 2-sided [-6.241 to 4.311], Standard Error of Mean 2.6535

9. Secondary Outcome: Change From Baseline of Cerebrospinal Fluid (CSF) Concentrations of Amyloid Beta (Aβ)
Description: CSF biomarker concentrations were analyzed for Aβ 1-40 and Aβ 1-42 using Innotest Enzyme-linked immunosorbent assays (ELISA) method. LS mean was derived using an ANCOVA model with fixed effects of baseline CSF, treatment, APOE4 Carrier Status (yes/no) and age at baseline.
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: nanograms per liter (ng/L)
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 51 | 54
nanograms per liter (ng/L)
  CSF Amyloid Beta 1-40 Modified ELISA - INNOTEST | 12151.386 (711.6120) | -587.063 (691.2989)
  CSF Amyloid Beta 1-42 Mod Modified ELISA - INNOTEST: number analyzed (Participants) | 51 | 52
  CSF Amyloid Beta 1-42 Mod Modified ELISA - INNOTEST | 1045.570 (42.6843) | 49.160 (42.2627)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Cerebrospinal Fluid Amyloid Beta 1-40 Modified ELISA - INNOTEST; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = 12738.449, 95% CI 2-sided [10757.047 to 14719.851], Standard Error of Mean 998.7048
Statistical Analysis 2: Comparison: Solanezumab vs Placebo; Cerebrospinal Fluid Amyloid Beta 1-42 Mod Modified ELISA - INNOTEST; Test type: Superiority; p < 0.001, ANCOVA — p-value using ANCOVA model for endpoint measures: CHG = Baseline + APOE4 + AGE + Treatment; LS Mean difference (Final Values) = 996.411, 95% CI 2-sided [875.873 to 1116.948], Standard Error of Mean 60.7404

10. Secondary Outcome: Change From Baseline in Brain Volume as Measured by Volumetric Magnetic Resonance Imaging (vMRI)
Description: Alzheimer's disease is also associated with pronounced brain atrophy, reflecting bulk neurodegenerative loss of gray and white matter. Progression of brain atrophy is assessed by vMRI, providing regional quantification of volume loss. Negative change from baseline indicates greater disease severity. Total hippocampal volume and Total Lateral Ventricular Volume were analyzed for vMRI parameters. LS mean was derived using an ANCOVA model with fixed effects of baseline vMRI value, treatment, age at baseline, education, APOE4 Carrier Status (yes/no), and baseline florbetapir cortical SUVr.
Time Frame: Baseline, Week approximately 240
Population: All randomized participants who have a baseline score and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: cubic centimeter (cm^3)
Arm/Group | Solanezumab | Placebo
Number analyzed (Participants) | 561 | 578
cubic centimeter (cm^3)
  Total hippocampal volume | -0.369 (0.0276) | -0.314 (0.0272)
  Total Lateral Ventricular Volume | 9.329 (0.3215) | 8.978 (0.3167)
Statistical Analysis 1: Comparison: Solanezumab vs Placebo; Total hippocampal volume; Test type: Superiority; p = 0.161, ANCOVA; LS Mean difference (Final Values) = -0.054, 95% CI 2-sided [-0.131 to 0.022], Standard Error of Mean 0.0388
Statistical Analysis 2: Comparison: Solanezumab vs Placebo; Total Lateral Ventricular Volume; Test type: Superiority; p = 0.437, ANCOVA; LS Mean difference (Final Values) = 0.351, 95% CI 2-sided [-0.535 to 1.236], Standard Error of Mean 0.4513

11. Secondary Outcome: Change From Baseline on the Clinical Dementia Rating-Sum of Boxes Score (CDR-SB)
Description: The CDR-SB is an interviewer administered scale and impairment is scored in each of categories: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 6 individual category ratings, or "box scores", were added together to give the CDR-Sum of Boxes which ranges from 0-18. Higher score indicates severe impairment.
Time Frame: Baseline, Week 336
Population: as for outcome 2
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline on the Computerized Cognitive Composite (C3)
Description: The C3 includes tasks from the CogState battery aimed at measuring processing speed, working memory, visual navigation, and executive function. The C3 also include 2 investigator-developed sensitive episodic memory probes of hippocampal function. A composite score is generated and CogState scores are measured on a linear scale (with no maximum score) and a reduction in scores compared to baseline indicates an improvement in cognitive functions.
Time Frame: Baseline, Week 336
Population: as for outcome 2
Arm/Group | Solanezumab/Solanezumab | Placebo/Solanezumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Double-blind (Placebo Controlled) Period (Baseline Up to Week 240); Open-label Extension Period (Week 240 Up to Week 444)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Solanezumab: Double-blind (Placebo Controlled) Period: Participants received 400 mg solanezumab followed by 800 mg solanezumab and then 1600 milligram solanezumab administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
- Placebo: Double-blind (Placebo Controlled) Period: Participants received placebo administered IV Q4W for approximately 240 weeks in double-blind (placebo-controlled) period.
- Solanezumab/Solanezumab: Open-label Extension Period: Participants who received solanezumab in double-blind period were administered 1600 mg solanezumab IV Q4W for 204 weeks (from week 240 to week 444) in open-label extension period.
- Placebo/Solanezumab: Open-label Extension Period: Participants who received placebo in double-blind period were administered 1600 mg solanezumab IV Q4W for 204 weeks (from week 240 to week 444) in open-label extension period.
Arm/Group | Solanezumab: Double-blind (Placebo Controlled) Period | Placebo: Double-blind (Placebo Controlled) Period | Solanezumab/Solanezumab: Open-label Extension Period | Placebo/Solanezumab: Open-label Extension Period
All-Cause Mortality (participants affected / at risk) | 6/572 | 7/591 | 7/383 | 5/401
Serious Adverse Events (participants affected / at risk) | 171/572 | 156/591 | 51/383 | 70/401
Other Adverse Events (participants affected / at risk) | 531/572 | 554/591 | 286/383 | 310/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Solanezumab: Double-blind (Placebo Controlled) Period (N=572) | Placebo: Double-blind (Placebo Controlled) Period (N=591) | Solanezumab/Solanezumab: Open-label Extension Period (N=383) | Placebo/Solanezumab: Open-label Extension Period (N=401)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node rupture (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (4) | 4 (4) | 3 (3) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 9 (9) | 9 (11) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brash syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (4) | 1 (2) | 2 (2) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 7 (7) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Medical device site photosensitivity reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst ruptured (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess of salivary gland (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ear infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1/238 (1) | 0/234 (0) | 0/162 (0) | 0/163 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 9 (9) | 0 (0) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rocky mountain spotted fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Central cord syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 6 (6) | 5 (6) | 5 (5)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 3 (3)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest x-ray abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (8) | 0 (0) | 6 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dedifferentiated liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/334 (1) | 0/357 (0) | 0/221 (0) | 0/238 (0)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/334 (0) | 1/357 (1) | 0/221 (0) | 0/238 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/238 (6) | 1/234 (1) | 1/162 (1) | 0/163 (0)
Prostate cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/238 (0) | 1/234 (1) | 0/162 (0) | 0/163 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Superficial siderosis of central nervous system (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 3 (3) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 4 (5) | 4 (4) | 0 (0) | 1 (1)
Vith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3/238 (3) | 0/234 (0) | 1/162 (1) | 1/163 (1)
Prostatitis (Reproductive system and breast disorders) | 1/238 (1) | 1/234 (1) | 0/162 (0) | 0/163 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Closed fracture manipulation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1/238 (1) | 0/234 (0) | 0/162 (0) | 0/163 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Solanezumab: Double-blind (Placebo Controlled) Period (N=572) | Placebo: Double-blind (Placebo Controlled) Period (N=591) | Solanezumab/Solanezumab: Open-label Extension Period (N=383) | Placebo/Solanezumab: Open-label Extension Period (N=401)
Atrial fibrillation (Cardiac disorders) | 19 (19) | 24 (27) | 5 (5) | 9 (12)
Tinnitus (Ear and labyrinth disorders) | 9 (9) | 20 (20) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 33 (35) | 27 (29) | 11 (13) | 5 (5)
Cataract (Eye disorders) | 61 (82) | 74 (99) | 18 (21) | 24 (30)
Abdominal discomfort (Gastrointestinal disorders) | 18 (20) | 12 (14) | 5 (5) | 5 (5)
Constipation (Gastrointestinal disorders) | 26 (28) | 18 (19) | 6 (6) | 10 (10)
Dental caries (Gastrointestinal disorders) | 14 (18) | 21 (24) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 78 (91) | 78 (99) | 17 (17) | 18 (19)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 31 (33) | 38 (40) | 9 (9) | 8 (8)
Nausea (Gastrointestinal disorders) | 33 (36) | 31 (33) | 11 (15) | 4 (4)
Chest pain (General disorders) | 21 (22) | 15 (15) | 7 (8) | 5 (5)
Fatigue (General disorders) | 56 (72) | 45 (52) | 7 (7) | 7 (7)
Oedema peripheral (General disorders) | 23 (26) | 19 (19) | 6 (6) | 2 (2)
Seasonal allergy (Immune system disorders) | 29 (31) | 24 (26) | 5 (5) | 3 (3)
Bronchitis (Infections and infestations) | 50 (61) | 62 (72) | 11 (11) | 8 (9)
Cellulitis (Infections and infestations) | 27 (35) | 27 (30) | 6 (6) | 6 (7)
Conjunctivitis (Infections and infestations) | 11 (14) | 20 (24) | 6 (6) | 1 (1)
Covid-19 (Infections and infestations) | 22 (22) | 22 (22) | 105 (111) | 108 (113)
Gastroenteritis (Infections and infestations) | 23 (23) | 21 (26) | 2 (2) | 5 (5)
Herpes zoster (Infections and infestations) | 19 (21) | 24 (25) | 6 (6) | 3 (3)
Influenza (Infections and infestations) | 49 (53) | 42 (47) | 4 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 117 (172) | 121 (183) | 12 (12) | 17 (18)
Pneumonia (Infections and infestations) | 23 (24) | 26 (28) | 3 (3) | 11 (11)
Sinusitis (Infections and infestations) | 59 (78) | 74 (94) | 14 (16) | 9 (10)
Tooth abscess (Infections and infestations) | 14 (16) | 26 (32) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 16 (17) | 18 (21) | 4 (4) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 174 (298) | 198 (348) | 41 (50) | 46 (54)
Urinary tract infection (Infections and infestations) | 82 (149) | 92 (139) | 34 (49) | 35 (50)
Viral upper respiratory tract infection (Infections and infestations) | 27 (33) | 39 (50) | 3 (3) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 21 (26) | 30 (32) | 3 (3) | 8 (9)
Contusion (Injury, poisoning and procedural complications) | 59 (77) | 56 (64) | 10 (11) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 170 (266) | 156 (278) | 66 (90) | 71 (95)
Ligament sprain (Injury, poisoning and procedural complications) | 31 (34) | 40 (43) | 6 (6) | 7 (7)
Meniscus injury (Injury, poisoning and procedural complications) | 18 (19) | 18 (20) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 43 (46) | 37 (39) | 9 (11) | 8 (9)
Skin abrasion (Injury, poisoning and procedural complications) | 34 (42) | 28 (36) | 3 (3) | 5 (6)
Skin laceration (Injury, poisoning and procedural complications) | 41 (44) | 53 (59) | 11 (12) | 14 (20)
Tooth fracture (Injury, poisoning and procedural complications) | 15 (16) | 28 (32) | 1 (1) | 5 (5)
Vaccination complication (Injury, poisoning and procedural complications) | 7 (9) | 14 (15) | 12 (12) | 5 (9)
Blood creatine phosphokinase increased (Investigations) | 14 (15) | 20 (20) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 (13) | 18 (19) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 114 (153) | 117 (153) | 39 (45) | 35 (41)
Arthritis (Musculoskeletal and connective tissue disorders) | 34 (37) | 34 (37) | 6 (6) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 77 (88) | 78 (90) | 23 (23) | 14 (14)
Bursitis (Musculoskeletal and connective tissue disorders) | 19 (19) | 24 (27) | 5 (5) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 39 (44) | 32 (34) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (32) | 22 (23) | 6 (6) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 25 (25) | 20 (21) | 1 (1) | 8 (8)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 50 (55) | 57 (66) | 13 (16) | 12 (13)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 20 (20) | 21 (21) | 5 (5) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 (56) | 53 (64) | 19 (20) | 13 (14)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 21 (22) | 17 (17) | 5 (5) | 9 (12)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 47 (71) | 53 (90) | 13 (15) | 17 (33)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (39) | 29 (53) | 19 (22) | 9 (19)
Balance disorder (Nervous system disorders) | 15 (16) | 19 (21) | 5 (7) | 2 (2)
Cerebral microhaemorrhage (Nervous system disorders) | 23 (27) | 41 (51) | 6 (8) | 11 (13)
Cognitive disorder (Nervous system disorders) | 50 (50) | 33 (33) | 10 (10) | 18 (18)
Dizziness (Nervous system disorders) | 79 (95) | 62 (72) | 19 (21) | 15 (20)
Headache (Nervous system disorders) | 112 (158) | 118 (157) | 22 (24) | 24 (27)
Memory impairment (Nervous system disorders) | 23 (23) | 16 (18) | 2 (2) | 4 (4)
Paraesthesia (Nervous system disorders) | 18 (20) | 25 (32) | 5 (5) | 4 (4)
Sciatica (Nervous system disorders) | 32 (39) | 21 (25) | 4 (5) | 4 (4)
Anxiety (Psychiatric disorders) | 38 (40) | 33 (33) | 17 (18) | 10 (11)
Depression (Psychiatric disorders) | 35 (35) | 38 (40) | 6 (6) | 9 (9)
Insomnia (Psychiatric disorders) | 34 (36) | 36 (37) | 8 (8) | 13 (14)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 14/238 (16) | 13/234 (13) | 4/162 (4) | 7/163 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (50) | 50 (60) | 9 (9) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 21 (23) | 3 (3) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 19 (21) | 4 (4) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 26 (35) | 28 (31) | 5 (8) | 6 (6)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 29 (34) | 26 (34) | 6 (6) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (19) | 24 (27) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 56 (63) | 39 (49) | 12 (15) | 9 (10)
Hypertension (Vascular disorders) | 58 (63) | 59 (61) | 17 (17) | 16 (18)

LIMITATIONS AND CAVEATS:
Per protocol and SAP, delayed-start analyses were not conducted because no treatment difference was observed at the end of the double-blind (placebo-controlled) period. Hence, data were not evaluated for outcome measure analyses (week 336), but safety data were analyzed for open-label extension period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT02008357/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02008357/SAP_001.pdf